CLINICAL TRIAL: NCT05904808
Title: Diuresis Efficacy in Ambulatory Chronic Heart Failure Patients With Volume Overload- Intra -Patient Comparison of Three Diuretics Regimens
Brief Title: The Heart Failure Diuresis Efficacy Comparison (DEA-HF) Study
Acronym: DEA-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Aharon (Ronnie) Abbo MD, Deputy Director, Cardio Vascular Research and Innovation Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0067-23-RMB
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Heart Failure; Diuretics Drug Reactions; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Acetazolamide; magnesium citrate

STUDY DESIGN:
Intervention Model Description: Single-site, single-arm, open-label, cross-over controlled study Randomization will determine the sequence of the three (3) regimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diuretic comparison (Active Comparator): each participant will be followed for 4 consecutive weeks. during which 3 different diuretic regimens will be given (random sequence). Last week follow up without protocol regimen.
  Interventions: Drug: IV Furosemide; Drug: IV Furosemide and PO Metolazone; Drug: IV Furosemide and IV Acetazolamide

INTERVENTIONS:
Drug: IV Furosemide — Given over 4-hour drip using IV pump, 40mg of the 250mg will be given as a bolus
Drug: IV Furosemide and PO Metolazone — Given over 4-hour drip using IV pump, 40mg of the 250mg will be given as a bolus +5mg PO Metolazone
Drug: IV Furosemide and IV Acetazolamide — Furosemide would be given over 4-hour drip using IV pump, 40mg of the 250mg will be given as a bolus.
  500mg IV Acetazolamide would be given in 100cc of saline over half an hour
  Other Names: Oral Magnesium citrate 600mg

SUMMARY:
To investigate the effectiveness of three (3) IV diuretic regimens to increase natriuresis in volume-overloaded HF patients, allowing for better decongestion and potentially resulting in improved clinical and biochemical parameters outcome.

DETAILED DESCRIPTION:
The study will assess the efficacy and safety of three (3) different clinically prevailing diuretic regimens. All three regimens are based on furosemide, as mentioned above- a 1st line HF GL2,3 recommended and MOH registered 7 for fluid decongestion, and the two adjuvants medications are also approved as diuretics in HF patients. Better natriuresis will lead to better decongestion in CHF patients with volume overload. It is expected that the better natriuresis will lead to better decongestion, and improvement in favorable markers parameters such as NT pro BNP.

The trial will investigate treatment regimens, readily available, clinically approved ("on-label" in Israel), which can be very easily administered, through an IV infusion or IV and PO administration without additional extra testing or invasive monitoring. The setting is in an established dedicated HF day-care unit at the cardiology department of Rambam Health Campus (RMC)- a tertiary referral academic center.

The knowledge gathered in this study, could be easily adopted by every clinic or hospital in a quick manner with considerable cost-savings with regards to health care expenditure.

Importantly, this study will examine which application of existing decongestive therapies (not novel drugs), based on strong scientific reasoning, will result in a better outcome for patients. Therefore, data from the study will provide information regarding the safety and efficacy of diuretic treatment in the above-mentioned patient population.

The study intends to be a real-life study, in the manner of:

1. Conducted in an established, protocol-operated setting
2. Essential only recruitment restrictions
3. Without any additional testing to the day care standard of care
4. Have minimal or no additional expected risk for the patient (comparison between standard diuretic regimens)
5. Have very clinically meaningful endpoints.

Therefore, this study should be considered a 'Low-intervention clinical trial' as:

1. The investigational medicinal products, which are used in clinical practice and approved, have a very low-risk profile and are well-known to general cardiologists and internists worldwide.
2. According to the protocol of the clinical trial, all investigational medicinal products will be used in accordance with EU and US marketing approval according to published guidelines. Note: from commercial and supply chain reasons oral metolazone and IV acetazolamide are imported by medical institutions in Israel by means of group "29 gimel" form. Both are FDA and EU labeled for HF treatment.
3. No additional diagnostic or monitoring procedures are asked. Hence, minimal additional risk or burden to the safety of the subjects compared to normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent must be obtained before any study assessment is performed.
2. Male or female patients 18 years of age or older
3. Confirmed Diagnosis of Heart Failure (per ESC guidelines 20212)
4. At least one sign of active congestion at recruitment: Jugular venous pressure(JVP)/Ascites/Edema/Pulmonary rales/Pleural effusion/ Lung ultrasound B lines >3 lines (at 6 sites).
5. Patient is at least on two heart failure drugs including: BB, MRA, sGLT2i, ACEI/ARB/ARNI (or has a clinical reason for its absence) and on oral diuretics for the last 30 days before study inclusion.

Exclusion Criteria:

1. History of myocardial infraction in the last 14 days prior to patient randomization.
2. History of a cardiac transplantation and/or ventricular assist device.
3. Mean blood pressure <60 mmHg at screening
4. Simultaneous use of intravenous inotropes, vasopressors or nitroprusside due to acute decompensated heart failure in the last 14 days.
5. Estimated glomerular filtration rate <20ml/min/1.73m2 at screening
6. Any circumstances where urine collection is not possible.
7. Use of renal replacement therapy or ultrafiltration 30 days prior to patient randomization.
8. Subjects who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Sodium weight | 1st week visit (time zero)
  Na Weight (Spot Na * total volume of urine)
Sodium weight | 1 week after 1st visit
  Na Weight (Spot Na * total volume of urine)
Sodium weight | 2 weeks after 1st visit
  Na Weight (Spot Na * total volume of urine)

SECONDARY OUTCOMES:
Urine Volume | 1st week visit (time zero)
  Total urinary volume starting from initiation of intravenous (IV) therapy for 6 hours
Urine Volume | 1 week after 1st visit
  Total urinary volume starting from initiation of intravenous (IV) therapy for 6 hours
Urine Volume | 2 weeks after 1st visit
  Total urinary volume starting from initiation of intravenous (IV) therapy for 6 hours
Rate of symptomatic hypotension events | A week after 1st visit
  Systolic BP <90mmhg with symptoms
Rate of symptomatic hypotension events | 2 weeks after 1st visit
  Systolic BP <90mmhg with symptoms
Rate of symptomatic hypotension events | 3 weeks after 1st visit
  Systolic BP <90mmhg with symptoms
rate of worsening renal function events | A week after 1st visit
  WRF defined as a >0.3 mg/dL increase in serum Cr, or a >20% decrease in eGFR by the CKDEPI formula
rate of worsening renal function events | 2 weeks After 1st visit
  WRF defined as a >0.3 mg/dL increase in serum Cr, or a >20% decrease in eGFR by the CKDEPI formula
rate of worsening renal function events | 3 weeks after 1st visit
  WRF defined as a >0.3 mg/dL increase in serum Cr, or a >20% decrease in eGFR by the CKDEPI formula
Rate of hyponatremia during treatment phase | A week after 1st visit
  Hyponatremia <133mmol/dl
Rate of hyponatremia during treatment phase | 2 weeks after 1st visit
  Hyponatremia <133mmol/dl
Rate of hyponatremia during treatment phase | 3 weeks after 1st visit
  Hyponatremia <133mmol/dl
Rate of dyskalemia events during treatment phase | A week after 1st visit
  Dyskalemia defined as <3.5 or >5.6mmol/dl
Rate of dyskalemia events during treatment phase | 2 weeks after 1st visit
  Dyskalemia defined as <3.5 or >5.6mmol/dl
Rate of dyskalemia events during treatment phase | 3 weeks after 1st visit
  Dyskalemia defined as <3.5 or >5.6mmol/dl
Rate of metabolic acidosis events requiring NaHCO3 supplements | A week after 1st visit
  Rate of Metabolic acidosis (requiring NaHCO3 supplements) events
Rate of metabolic acidosis events requiring NaHCO3 supplements | 2 weeks after 1st visit
  Rate of Metabolic acidosis (requiring NaHCO3 supplements) events
Rate of metabolic acidosis events requiring NaHCO3 supplements | 3 weeks after 1st visit
  Rate of Metabolic acidosis (requiring NaHCO3 supplements) events

OTHER OUTCOMES:
Change in plasma volume | A week after 1st visit
  Assessed using weight and HCT
Change in plasma volume | 2 weeks after 1st visit
  Assessed using weight and HCT
Change in plasma volume | 3 weeks after 1st visit
  Assessed using weight and HCT
Rate of magnesium deficiency a week after treatment | A week after 1st visit
  Defined as Mag levels <1.6mmol/dl
Rate of magnesium deficiency a week after treatment | 2 weeks after 1st visit
  Defined as Mag levels <1.6mmol/dl
Rate of magnesium deficiency a week after treatment | 3 weeks after 1st visit
  Defined as Mag levels <1.6mmol/dl
Change in body weight a week after each IV regimen | A week after 1st visit
  weight scale
Change in body weight a week after each IV regimen | 2 weeks after 1st visit
  weight scale
Change in body weight a week after each IV regimen | 3 weeks after 1st visit
  weight scale
Change in BNP level a week after each IV treatment | A week after 1st visit
  Plasma Nt-ProBNP
Change in BNP level a week after each IV treatment | 2 weeks after 1st visit
  Plasma Nt-ProBNP
Change in BNP level a week after each IV treatment | 3 weeks after 1st visit
  Plasma Nt-ProBNP
Change in decongestion achieved by change in congestion score- week after treatment | A week after 1st visit
  A composite score of: pedal edema, orthopnea, ultrasound evidence of pleural effusion, ascites and B-lines. each getting a rank between 0-4. total score can range from 0-16, where higher score indicates worse congestion and prognosis status.
Change in decongestion achieved by change in congestion score- week after treatment | 2 weeks after 1st visit
  A composite score of: pedal edema, orthopnea, ultrasound evidence of pleural effusion, ascites and B-lines. each getting a rank between 0-4. total score can range from 0-16, where higher score indicates worse congestion and prognosis status.
Change in decongestion achieved by change in congestion score- week after treatment | 3 weeks after 1st visit
  A composite score of: pedal edema, orthopnea, ultrasound evidence of pleural effusion, ascites and B-lines. each getting a rank between 0-4. total score can range from 0-16, where higher score indicates worse congestion and prognosis status.

CONTACTS AND LOCATIONS:
Overall Officials: Aharon Abbo, MD, Principal Investigator — Rambam
Locations (1):
- Rambam MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT05904808/SAP_000.pdf